CLINICAL TRIAL: NCT02222857
Title: Prophylactic Laser Photocoagulation and Vitrectomy for Acute Retinal Necrosis
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201406118RIND
Record Dates: First submitted 2014-08-20; First posted 2014-08-21 (Estimated); Last update posted 2018-04-26 (Actual); Status verified 2014-08

CONDITIONS: Acute Retinal Necrosis; Retinal Detachment; Laser Photocoagulation; Vitrectomy
Keywords: Acute retinal necrosis; Retinal detachment; Laser photocoagulation; Vitrectomy
MeSH Terms: conditions — Retinal Necrosis Syndrome, Acute; Retinal Detachment

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Acute retinal necrosis (ARN) is a rare infectious retinitis which can potentially lead to devastating visual outcomes. ARN is diagnosed on the basis of the clinical appearance and disease course according to the diagnostic criteria proposed by the American Uveitis Society: (1) one or more foci of retinal necrosis with discrete borders in the peripheral retina; (2) rapid progression in the absence of antiviral therapy; (3) circumferential spread; (4) occlusive vasculopathy with arteriolar involvement; and (5) a prominent inflammatory reaction in the vitreous and anterior chambers.

Herpesvirus infection, especially varicella-zoster virus (VZV) and herpes simplex virus (HSV), was presumed to be the pathogenic agent in the pathogenesis of ARN. Medical treatment with systemic antiviral agent had been the base of the therapy of ARN for decades and such treatment usually result in regression of retinitis.

However, the visual outcome of ARN remains poor. The major causes of poor visual prognosis in ARN are retinal detachment and optic nerve or macular involvement by ischemic vasculopathy. Less frequent causes include macular hole formation, macular pucker, or hypotony. Rhegmatogenous retinal detachment may occur in 75 % of the untreated eyes. It may occur weeks to months after the onset of inflammation due to delayed formation of retinal breaks, which result from the combination of necrotic retina and vitreoretinal traction.

Therefore, application of argon laser retinopexy prophylactically posterior to necrotic retina or prophylactic vitrectomy to reduce inflammatory factors and the vitreoretinal traction had been used to protect the healthy area from detachment. However, the results were varied and there is no consensus on the efficacy and indications of those prophylactic procedures. We had applied the prophylactic procedure in our treatment for ARN. We aim to access the efficacy of the treatment strategy of ARN and the correlated factors to the outcomes.

DETAILED DESCRIPTION:
Between 1995 and 2013, the charts of 20 patients (21 eyes) with a clinical diagnosis of ARN and a complete ophthalmic examination at National Taiwan University Hospital were reviewed. The study was approved by the Ethics Committee and Institutional Review Board of National Taiwan University Hospital.

The clinical data recorded included patient demographics, refractive error, lens status, best corrected visual acuity (BCVA), all treatments and retinal anatomical status. Visual acuities and examination findings were recorded at presentation and subsequent follow-up periods for at least 6 months. The area of retina involved was determined by review of retinal drawings and fundus photos by single reader.

All the patients were admitted for intravenous injection of Acyclovir (30mg/kg/day, in 3 divided doses) for 10-14 days and then shifted to oral Acyclovir (30mg/kg/day) at least for further 10-14 days. Systemic corticosteroid and Aspirin were also given. Prophylactic laser photocoagulation was arranged on normal retina to surround the posterior edge of the active lesions if the media was clear enough to approach. If vitritis persisted without improvement under systemic antiviral agent or retinal detachment was noted, vitrectomy would be performed. Visual acuities and retinal anatomical results were recorded during follow-up after procedures. The visual acuity was converted to logarithm of the minimum angle of resolution (logMAR) values for statistical analysis.

Statistical analysis The continuous values are expressed as means ± standard deviation (SD). The differences among the continuous variables were assessed using the Mann-Whitney U test. Non-continuous variables were analyzed by Fisher's exact test. The level of statistical significance was set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

●Patients with clinical diagnosis of acute retinal necrosis.

Exclusion Criteria:

* Patients with history of retinal detachment.
* Patients with history of other causes of severe retinal atrophy or necrosis.
* HIV positive patients.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute retinal necrosis
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2014-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Best-corrected visual acuity | 1 year
  Best-corrected visual acuity during follow up and its correlated factors

SECONDARY OUTCOMES:
Retinal status | 1 year
  Retinal status by ophthalmoscopy to see the incidence of retinal detachment and its correlated factors

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Ping Lin, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan